CLINICAL TRIAL: NCT04811378
Title: Randomised Controlled Trial: HaemoCerTM Versus no HaemoCerTM in Breast Cancer Surgery to Reduce Postoperative Drainage Output
Brief Title: HaemoCerTM Application in Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christian Singer, Univ.-Prof. Dr.med.univ. MPH, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1178/2017
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Breast Neoplasm Female; Mastectomy, Segmental

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HaemoCer (Active Comparator)
  Interventions: Other: HaemoCer
- No HaemoCer (No Intervention)

INTERVENTIONS:
Other: HaemoCer — Randomized application of 3g haemostatic powder (HaemoCer) in the wound site during breast-conserving surgery.
  Arms: HaemoCer

SUMMARY:
HaemoCer is a hemostatic agent to control bleedings during surgical procedures by accelerating natural hemostasis and is frequently applied during breast conserving surgery in women with breast cancer. There is however no adequate data available on the efficacy of HaemoCer regarding seroma formation or drainage output. The objective of this study is to investigate whether the intraoperative application of haemostatic powder (HaemoCer) in breast-conserving surgery in breast cancer patients reduces the postoperative drainage output and number of days until drain removal (number of hospitalization days).

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer undergoing breast-conserving surgery
* No previous breast-conserving surgery on the same site
* ≥ 18 years age
* no current pregnancy
* Informed consent

Exclusion Criteria:

Patients with previous breast-conserving surgery on the same site

-

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Total volume of postoperative drained fluid (per breast) | 7 days
Number of days until drain removal (n) | 7 days

SECONDARY OUTCOMES:
Total volume of postoperative drained fluid from the axillary fossa in case of axilla surgery (sentinel lymphonodectomy, axillary dissection) | 7 days
Rate of immediate postoperative infection on the breast surgery site | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Singer, Prof., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria